CLINICAL TRIAL: NCT00219063
Title: A 26 Week, Double-blind, Randomized, Multicenter, Parallel Group, Active-controlled Study Comparing Aliskiren to Ramipril With Optional Addition of Hydrochlorothiazide, Followed by a 4 Week Double-blind, Randomized, Placebo-controlled Withdrawal in Patients With Essential Hypertension
Brief Title: A Clinical Study to Compare an Aliskiren Based Hypertensive Regimen With a Ramipril Based One Followed by a Randomized Withdrawal.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2306
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Hypertension
Keywords: Hypertension, aliskiren, blood pressure, Ramipril, hydrochlorothiazide
MeSH Terms: conditions — Hypertension | interventions — aliskiren

INTERVENTIONS:
Drug: aliskiren

SUMMARY:
To compare the aliskiren regimen versus the ramipril regimen on reduction in Blood Pressure.

ELIGIBILITY:
Inclusion Criteria

* Patients with essential hypertension
* Patients who are eligible and able to participate in the study

Exclusion Criteria

* Severe hypertension
* History or evidence of a secondary form of hypertension
* History of Hypertensive encephalopathy or cerebrovascular accident. Other protocol-defined inclusion exclusion criteria also apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 844 (Actual)
Dates: Start 2005-02; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in diastolic blood pressure after 26 weeks

SECONDARY OUTCOMES:
Change from baseline in systolic blood pressure after 26 weeks
Change from baseline in diastolic blood pressure after 6 weeks and 12 weeks
Change from baseline in systolic blood pressure after 6 weeks and 12 weeks
Blood pressure control target of < 140/90 mmHg after 6, 12, and 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States

REFERENCES:
- [Result] Andersen K, Weinberger MH, Egan B, Constance CM, Ali MA, Jin J, Keefe DL. Comparative efficacy and safety of aliskiren, an oral direct renin inhibitor, and ramipril in hypertension: a 6-month, randomized, double-blind trial. J Hypertens. 2008 Mar;26(3):589-99. doi: 10.1097/HJH.0b013e3282f3ad9a. PMID 18300872